CLINICAL TRIAL: NCT05758532
Title: Harnessing the Beneficial Non-specific Effects of Measles-mumps-rubella Vaccine in Children on Infection With Unrelated Pathogens and Allergic Diseases - a Single-centre Phase IV RCT With a Factorial Design
Brief Title: Non-specific Effects of a Modified Measles Vaccination Schedule to Prevent Allergy and Unrelated Infection in Children
Acronym: NEMAU
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Laure Pittet, MD-PhD (Other)
Responsible Party: Sponsor-Investigator, Laure Pittet, MD-PhD, Clinical Scientist, Pediatric Clinical Research Platform
Organization: Pediatric Clinical Research Platform (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2022-00616; Ambizione n° PZ00P3_209050 (Other Grant/Funding Number: Swiss National Science Foundation); STARTER-MD n° RS08-08 (Other Grant/Funding Number: Foundation Louis-Jeantet and Private Foundation of the HUG); PRD n° 4-2022-I (Other Grant/Funding Number: University Hospitals of Geneva)
Record Dates: First submitted 2023-02-10; First posted 2023-03-07 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Tract Infections; Infections; Allergy; Eczema
Keywords: Non-specific/off-target effect of vaccine
MeSH Terms: conditions — Respiratory Tract Infections; Infections; Hypersensitivity; Eczema | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Intervention Model Description: Phase IV, single-centre, 4-group, open-label, randomised controlled trial with a factorial design (primary outcome analysed as a 2-group trial)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C.C. : Both MMR doses given on current schedule (9 months and 12 months) (Active Comparator): Measles-mumps-rubella (MMR) vaccine 0.5 ml injected intramuscularly, at:
  * 9 months (= current Swiss schedule)
  * 12 months, concomitant with other vaccines (= current Swiss schedule)
  Interventions: Biological: Measles-Mumps-Rubella vaccine (MMR)
- M.C. : 1st MMR on modified schedule (6 months) and 2nd MMR on current schedule (12 months) (Experimental): Measles-mumps-rubella (MMR) vaccine 0.5 ml injected intramuscularly, at:
  * 6 months (= modified schedule)
  * 12 months, concomitant with other vaccines (= current Swiss schedule)
  Interventions: Biological: Measles-Mumps-Rubella vaccine (MMR)
- C. M. : 1st MMR on current schedule (9 months) and 2nd MMR on modified schedule (13 months) (Experimental): Measles-mumps-rubella (MMR) vaccine 0.5 ml injected intramuscularly, at:
  * 9 months (= current Swiss schedule)
  * 13 months, distant from other vaccines (= modified schedule)
  Interventions: Biological: Measles-Mumps-Rubella vaccine (MMR)
- M.M. : Both MMR doses given on modified schedule (6 months and 13 months) (Experimental): Measles-mumps-rubella (MMR) vaccine 0.5 ml injected intramuscularly, at:
  * 6 months (= modified schedule)
  * 13 months, distant from other vaccines (= modified schedule)
  Interventions: Biological: Measles-Mumps-Rubella vaccine (MMR)

INTERVENTIONS:
Biological: Measles-Mumps-Rubella vaccine (MMR) — 0.5 ml of MMR vaccine injected intramuscularly in the deltoid region or in the anterolateral area of the thigh

SUMMARY:
The goal of this clinical trial is to evaluate the off-target/non-specific effects of the measles-mumps-rubella (MMR) vaccine in children.

DETAILED DESCRIPTION:
The overall objective of this project is to assess, in a randomised control trial (RCT), the effects of a "modified" MMR schedule in children, by an in-depth characterisation of both the clinical effects and the underlying immunomodulatory changes.

The current Swiss administration schedule of giving MMR at 9 and 12 months of age ("current schedule") will be compared with a "modified schedule". This is expected to maximise the beneficial non-specific effects of MMR by giving it at 6 and 13 months of age, separately from other vaccines ("modified schedule"). Factorial analysis will enable assessment of the benefit of the intervention on each of the two doses of MMR separately or in combination.

The clinical aims are to determine whether a modified schedule of MMR administration reduces both the risk and severity of: (i) infections with unrelated pathogens and (ii) atopic and allergic diseases.

The laboratory aims are to: (i) quantify and characterise the immunological non-specific effects of MMR, and (ii) identify the biological pathways and molecular mechanisms that are altered by MMR vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by signature
2. 6-month-old children
3. In overall good health, without any clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.) and no clinically significant abnormal finding on history and/or physical examination
4. Fully immunised for age according to the Swiss vaccination schedule

   1. with at least 2 doses of DTP-containing vaccine
   2. the last dose of vaccine received at least 2 weeks prior to enrolment

Exclusion Criteria:

1. Contra-indications to MMR, including

   1. immunosuppression (i.e. proven, suspected, or planned)
   2. allergy to a component of the vaccine
   3. receipt of a live-attenuated vaccine in the four weeks prior to inclusion
2. Vaccine refusal
3. Indication for an early MMR vaccination, including

   1. Measles outbreak
   2. Planned immunosuppression (indication to an accelerated schedule to be completed before starting an immunosuppressive treatment)
   3. Travel to a region with a high risk of measles outbreak
4. Indication for vaccination with MMR-varicella (MMRV) instead of MMR, including

   1. severe eczema
   2. parental will
5. Parental inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, known/suspected non-compliance, substance abuse, etc.
6. Plan to move out of the country or have prolong absence during the trial
7. Other sibling included in the trial (in the case of multiple pregnancy, only one child can be randomised)
8. Any temporary contra-indication to MMR, including child being sick (active significant illness, inclusion can be delayed a few days until the illness resolves)

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Incidence of parent-reported respiratory infections between 6 months and 9 months of age using fortnightly REDCap questionnaires, with validation of data by confirmation with treating paediatrician and medical records.

SECONDARY OUTCOMES:
Infection: Time to first infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  For participants who have an event:
  Date of event onset - date of randomisation
  For participants who did not have an event:
  Earliest censoring date - date of randomisation
Infection: Time to first infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  For participants who have an event:
  Date of event onset - date of randomisation
  For participants who did not have an event:
  Earliest censoring date - date of randomisation
Infection: Prevalence of infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  number of participants who have an event / total number of participants
Infection: Prevalence of infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  number of participants who have an event / total number of participants
Infection: Incidence of infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  number of events / total time of follow-up
Infection: Incidence of infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  number of events / total time of follow-up
Infection: Number of days free of infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  number of days free of event / total days of follow-up of participants
Infection: Number of days free of infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  number of days free of event / total days of follow-up of participants
Infection severity: Duration of infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Per event, calculated as: date of recovery - date of onset
Infection severity: Duration of infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Per event, calculated as: date of recovery - date of onset
Infection severity: Antibiotic use for infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Per event, defined as a binary variable (yes/no)
Infection severity: Antibiotic use for infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Per event, defined as a binary variable (yes/no)
Infection severity: Hospitalisation for infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Per event, defined as a binary variable (yes/no)
Infection severity: Hospitalisation for infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Per event, defined as a binary variable (yes/no)
Infection severity: Outcome of infection within the 3 months following randomisation | Measured over the 3 months following randomisation
  Per event, defined as a categorical variable (uneventful/complication or sequel/death)
Infection severity: Outcome of infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Per event, defined as a categorical variable (uneventful/complication or sequel/death)
Incidence of respiratory infection within the 18 months following randomisation | Measured over the 18 months following randomisation
  Incidence of parent-reported respiratory infections between 6 months and 24 months of age using fortnightly REDCap questionnaires, with validation of data by confirmation with treating paediatrician and medical records.

OTHER OUTCOMES:
Allergic/atopic diseases: time to first allergic/atopic disease flare within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  For participants who have a flare:
  Date of event onset - date of randomisation
  For participants who did not have a flare:
  Earliest censoring date - date of randomisation
Allergic/atopic diseases: time to first allergic/atopic disease flare within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  For participants who have a flare:
  Date of event onset - date of randomisation
  For participants who did not have a flare:
  Earliest censoring date - date of randomisation
Allergic/atopic diseases: Prevalence of allergic/atopic disease within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  number of participants who have a flare / total number of participants
Allergic/atopic diseases: Prevalence of allergic/atopic disease within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  number of participants who have a flare / total number of participants
Allergic/atopic diseases: Incidence of allergic/atopic disease flare within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  number of flares / total time of follow-up
Allergic/atopic diseases: Incidence of allergic/atopic disease flare within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  number of flares / total time of follow-up
Allergic/atopic diseases: Days free of allergic/atopic disease flare within the 3 months following randomisation | Measured over the 3 months following randomisation
  Calculated as:
  number of days free of flare / total days of follow-up of participants
Allergic/atopic diseases: Days free of allergic/atopic disease flare within the 18 months following randomisation | Measured over the 18 months following randomisation
  Calculated as:
  number of days free of flare / total days of follow-up of participants
Eczema severity: Difference in eczema severity as assessed by SCORAD at 3 months following randomisation | Measured at 3 months after randomisation
  Calculated as the difference in SCORAD score
Eczema severity: Difference in eczema severity as assessed by SCORAD at 18 months following randomisation | Measured at 18 months after randomisation
  Calculated as the difference in SCORAD score
Eczema severity: Difference in eczema severity as assessed by POEM at 3 months following randomisation | Measured at 3 months after randomisation
  Calculated as the difference in POEM score
Eczema severity: Difference in eczema severity as assessed by POEM at 18 months following randomisation | Measured at 18 months after randomisation
  Calculated as the difference in POEM score
Eczema severity: Difference in eczema impact on quality of life at 3 months following randomisation | Measured at 3 months after randomisation
  Assessed by IDQOL score
Eczema severity: Difference in eczema impact on quality of life at 18 months following randomisation | Measured at 18 months after randomisation
  Assessed by IDQOL score
Eczema severity: Topical steroid use for eczema within 3 months following randomisation | Measured over the 3 months following randomisation
  Per event, defined as a binary variable (yes/no)
Eczema severity: Topical steroid use for eczema within the 18 months following randomisation | Measured over the 18 months following randomisation
  Per event, defined as a binary variable (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Laure F Pittet, MD-PhD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Under the terms of the funding agreement with the Swiss National Science Foundation, the NEMAU trial has a data sharing agreement in place.
  An anonymised Individual Participant Data (IPD) dataset and a data dictionary will be provided to a FAIR platform after database lock.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After database lock, a 12-month embargo period will be in place, to allow adequate time for analyses and publication outputs. Data transfer to a FAIR plateform will occur during the embargo period.
Access Criteria: Researchers from a recognised research institution can approach the PI for access of data.
  The researcher will need to provide evidence that the proposed use of the data has been ethically reviewed and approved by an Institutional Review Board (IRB)/ Human Research Ethics Committee(HREC), and accept HUG's conditions, under a collaborator agreement.